CLINICAL TRIAL: NCT03003429
Title: Correlation Study Between Heart Rate Variability and Anxiety in Anorexia Nervosa
Acronym: VARIASTRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0376; 2016-A01659-42 (Other: ID-RCB)
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Anorexia Nervosa
Keywords: Heart rate variability; anxiety; Autonomic dysfunction
MeSH Terms: conditions — Anorexia Nervosa; Anxiety Disorders; Primary Dysautonomias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart rate monitor (Experimental): The intervention consist in monitoring the heart rate variability during one night by using a heart rate monitor and a Polar RS800CX
  Interventions: Other: Heart rate monitor

INTERVENTIONS:
Other: Heart rate monitor — The intervention consist in monitoring the heart rate variability during one night by using a heart rate monitor and a Polar RS800CX

SUMMARY:
The heart rate variability (HRV) is a measure of the autonomic nervous system (ANS). In the model of anorexia nervosa, ANS is disturbed with mostly a predominance of activation of the parasympathetic nervous system and a decrease of the sympathetic system. Various explanations of this these dysfunctions are proposed in literature, mainly malnutrition, physical hyperactivity, anxiety, that are known characteristics of anorexia nervosa.

The primary aim of this study is to evaluate correlation between ANS dysfunction and anxiety in anorexia nervosa.

Other objectives of this study are firstly to evaluate correlation between ANS dysfunction and others parameters (weight, body mass index, depression, physical activity, purgative ou restrictive type, duration of disease, smoking) in anorexia nervosa and secondly to see if HRV is a predictive parameter of the evolution of anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged from 18 to 65 years
* Criteria of anorexia nervosa (DSM V)
* Body mass index (BMI) < 18 kg/m2
* Written consent to participate in the study
* Patient affiliated to a social security system

Exclusion Criteria:

* Pacemaker or other implantable electronic device
* Current comorbidity psychiatric disorder according to Axis I of DSM IV : severe depression (BDI > 8/13), substance use disorder .
* Psychotropic drugs or ongoing steroid therapy ;
* Pregnancy or breast-feeding ;
* History or known cardiovascular disorder, including hypertension ( > 140/90 mmHg ) , heart failure, arrhythmia and conduction disorder .
* Major protected by a legal protection
* Minors
* Patient involved in another research with an exclusion period ongoing at the run-in

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Statistical correlation between autonomic dysfunction (measured by HRV) and anxiety (measured by questionnaire) | at day 0
  The composite measure consists of the following :- Time and spectral-domain measures of HRV measured by nocturn registration with heart rate monitor and polar RS800CX Time domain - NN (normal-to-normal R-R interval), HRV index (total number of all NN/ the height of the histogram of all NN), SDNN (standard deviation of the NN), RMSSD (the root mean square of differences of successive NN), NN50 (Number of pairs of adjacent NN intervals differing by more than 50 ms in the entire recording) and pNN50 (NN50/total number of all NN), SDANN (Standard deviation of the average of NN intervals in all 5-minute segments of a long recording), SDNNIDX (Mean of the standard deviation in all 5-minute segments of a long recording) Frequency domain - VLF Power (very low frequency; <0.04 Hz), LF Power (low frequency; 0.04~0.15 Hz), HF Power (high frequency; 0.15~0.4 Hz), LF/HF ratio value
  - State-Trait Anxiety Inventory: version Y (STAI- form Y) - Morning blood cortisol level and serum prealbumin lev

SECONDARY OUTCOMES:
Statistical correlation between autonomic dysfunction (measured by HRV) and measures of Beck Depression inventory | at day 0
  Beck Depression inventory : Version 2 in french (BDI-II)
Statistical correlation between autonomic dysfunction (measured by HRV) and measures of Beck Depression inventory | at 6 months
  Beck Depression inventory : Version 2 in french (BDI-II)
Statistical correlation between autonomic dysfunction (measured by HRV) and measures of International physical activity questionnaire | at 6 months
  International physical activity questionnaire (IPAQ) - French version
Statistical correlation between autonomic dysfunction (measured by HRV) and measures of International physical activity questionnaire | at day 0
  International physical activity questionnaire (IPAQ) - French version

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain ICETA, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France